CLINICAL TRIAL: NCT07141225
Title: Application of the "Off-Clamp And Sutureless" Technique in Robot-Assisted Partial Nephrectomy: A Single-Center, Prospective Cohort Study
Brief Title: Application of the "Off-Clamp And Sutureless" Technique in Robot-Assisted Partial Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shao Pengfei (Other)
Responsible Party: Sponsor-Investigator, Shao Pengfei, Professor, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-568
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Renal and Urinary Disorders; Renal Cancer; Renal Particial
Keywords: robot-assisted partial nephrectomy; off-clamp; sutureless; postoperative renal function preservation
MeSH Terms: conditions — Urologic Diseases; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Off-Clamp Sutureless Group (Experimental)
  Interventions: Procedure: Off-Clamp Sutureless Technique

INTERVENTIONS:
Procedure: Off-Clamp Sutureless Technique — During the procedure, the renal artery and its branches are not clamped. The tumor is completely resected with a gross margin of 0.5-1 cm from its edge. Monopolar or bipolar electrocautery is used for hemostasis during resection. Following tumor removal, the renal resection bed is subjected to meticulous hemostasis, followed by the application of hemostatic agents without suture closure.

SUMMARY:
The detection rate of renal masses smaller than 7 cm has significantly increased in recent years. To preserve postoperative renal function to the greatest extent possible, guidelines from the European Association of Urology (EAU), the National Comprehensive Cancer Network (NCCN), and others have endorsed partial nephrectomy (PN) as the preferred treatment strategy for small renal masses.

In conventional PN, it is necessary to clamp the renal artery or its branch arteries and employ a double-layer suturing technique to close the resection bed. This controls bleeding, maintains a clear surgical field, and prevents postoperative urinary leakage. The maximum safe duration of warm ischemia to avoid irreversible renal parenchymal damage remains controversial, though most studies indicate a window of 20-30 minutes. Consequently, the "off-clamp sutureless" concept has gained prominence. Its core principle is to avoid renal artery clamping and replace suturing with novel haemostatic techniques, thereby maximizing the preservation of healthy renal parenchyma. With the diversification of haemostatic material options and the widespread adoption of robotic-assisted systems, the off-clamp sutureless strategy has become technically feasible for small renal masses with low complexity .

Multiple retrospective studies demonstrate that the off-clamp sutureless technique is non-inferior, offering safety and surgical outcomes comparable to conventional robot-assisted partial nephrectomy (RAPN). However, it is important to note that current research predominantly focuses on tumors ≤4 cm, is largely retrospective, and suffers from limited sample sizes. More robust, evidence-based medical evidence is required to support its application for larger tumors or those with complex anatomy.

DETAILED DESCRIPTION:
The detection rate of renal masses smaller than 7 cm has increased significantly in recent years. To maximize the preservation of postoperative renal function, guidelines from the European Association of Urology (EAU), the National Comprehensive Cancer Network (NCCN), and others have established partial nephrectomy (PN) as the preferred treatment option for small renal masses.

In conventional PN, the renal artery or its segmental branches must be clamped, and the renal defect is typically closed using a multilayer suturing technique to control bleeding, maintain a clear surgical field, and prevent postoperative urinary leakage. The maximum safe duration of warm ischemia time (WIT) remains controversial, though most studies suggest a limit of 20-30 minutes to avoid irreversible renal parenchymal damage. In murine models, renal damage increases steeply after ischemia exceeds 30 minutes. Furthermore, the renorrhaphy suture technique has a steep learning curve, and the suturing process itself can cause additional injury to the renal vasculature, potentially compromising global renal function . Notably, up to 30% of patients with normal preoperative renal function may experience a decline in their estimated glomerular filtration rate (eGFR) to <60 mL/min/1.73 m² post-surgery, and nearly 10% may suffer a >50% reduction in renal function . Consequently, the concept of a "zero-ischemia sutureless" approach has gained traction. Its core principle is to avoid renal artery clamping and replace suturing with novel haemostatic methods, thereby maximizing the preservation of healthy renal parenchyma. With the expanding array of haemostatic agents and the widespread adoption of robotic-assisted systems, the zero-ischemia sutureless strategy has become technically feasible for small renal masses with low complexity.

Findings from multiple retrospective studies indicate that the zero-ischemia sutureless technique is non-inferior, demonstrating comparable safety and surgical outcomes to standard robot-assisted partial nephrectomy (RAPN). A study by Antonio Franco et al. reported a median decline in overall renal function of only 10 mL/min after zero-ischemia sutureless surgery, supporting its role as a safe procedure that effectively preserves postoperative renal function and reduces complications. In a review, J. C. Moreno Cortés highlighted that replacing traditional artery clamping and suturing with mono- or bipolar electrocautery and new haemostatic agents offers a simpler and faster method for reconstruction. This approach simplifies the surgical steps without increasing the risk of complications. However, it is important to note that current research is predominantly focused on tumours ≤4 cm, is largely retrospective, and often involves small sample sizes. More robust evidence from prospective studies is needed to support the application of this technique for larger or anatomically complex tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old, regardless of gender;
2. Radiological findings demonstrating a tumor size of ≤7 cm;
3. Imaging studies showing no evidence of collecting system invasion;
4. Scheduled to undergo robot-assisted partial nephrectomy (RAPN).

Exclusion Criteria:

1. Preoperative imaging demonstrating evidence of distant metastasis or lymph node involvement;
2. Unilateral or bilateral multiple lesions not amenable to simultaneous resection;
3. History of prior systemic therapy, including molecular targeted therapy, immunotherapy, or chemotherapy;
4. Intraoperative conversion to radical nephrectomy;
5. Intraoperative conversion to open surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Bilateral Kidney GFR | 3 months after surgery
  Measured by 99mTc-DTPA

SECONDARY OUTCOMES:
Perioperative Complication Rate | 1 week after surgery
Intraoperative Blood Loss | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pengfei Shao, Professor, Principal Investigator — The First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), Nanjing, Jiangsu 210036
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Without obtaining prior consent from the participant.